CLINICAL TRIAL: NCT02070744
Title: A Phase 2, Randomized, Multicenter, Double Blind, Placebo Controlled Study to Evaluate Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics of VX-661 in Combination With Ivacaftor for 12 Weeks in Subjects With Cystic Fibrosis, Homozygous for the F508del CFTR Mutation With an Open-Label Extension
Brief Title: Study to Evaluate Safety and Efficacy of VX-661 in Combination With Ivacaftor in Subjects With Cystic Fibrosis, Homozygous for the F508del-CFTR Mutation With an Open-Label Expansion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VX13-661-103
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Cystic Fibrosis
Keywords: CF
MeSH Terms: conditions — Cystic Fibrosis | interventions — tezacaftor; ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- PC Phase: VX-661 50 mg q12h + IVA 150 mg q12h (Experimental): Participants received VX-661 50 milligram (mg) tablet plus Ivacaftor (IVA) 150 mg tablet every 12 hours (q12h) for 12 weeks.
  Interventions: Drug: VX-661; Drug: Ivacaftor
- PC Phase: VX 661 placebo q12h + IVA placebo q12h (Placebo Comparator): Participants received placebo matched to VX-661 tablet plus placebo matched to IVA tablet q12h for 12 weeks.
  Interventions: Drug: Placebo matched to VX-661; Drug: Placebo matched to Ivacaftor
- PC Phase: VX-661 100 mg qd + IVA 150 mg q12h (Experimental): Participants received two VX-661 50 mg tablets once daily (qd) plus IVA 150 mg tablet q12h for 12 weeks.
  Interventions: Drug: VX-661; Drug: Ivacaftor
- PC Phase: VX -661 placebo qd + IVA placebo q12h (Placebo Comparator): Participants received two placebo matched to VX-661 tablets qd plus placebo matched to IVA tablet q12h for 12 weeks.
  Interventions: Drug: Placebo matched to VX-661; Drug: Placebo matched to Ivacaftor
- OLE Phase: VX-661 100 mg qd + IVA 150 mg q12h (Experimental): Participants who completed 12 week PC phase underwent a washout period of at least 4 weeks before entering the OLE phase and received two VX-661 50 mg tablets qd plus IVA 150 mg tablet q12h for 48 weeks in OLE phase.
  Interventions: Drug: VX-661; Drug: Ivacaftor

INTERVENTIONS:
Drug: VX-661 — Tablet, oral use
  Arms: OLE Phase: VX-661 100 mg qd + IVA 150 mg q12h; PC Phase: VX-661 100 mg qd + IVA 150 mg q12h; PC Phase: VX-661 50 mg q12h + IVA 150 mg q12h
Drug: Ivacaftor — Film coated tablet, oral use
  Arms: OLE Phase: VX-661 100 mg qd + IVA 150 mg q12h; PC Phase: VX-661 100 mg qd + IVA 150 mg q12h; PC Phase: VX-661 50 mg q12h + IVA 150 mg q12h
Drug: Placebo matched to VX-661 — Tablet, oral use
  Arms: PC Phase: VX -661 placebo qd + IVA placebo q12h; PC Phase: VX 661 placebo q12h + IVA placebo q12h
Drug: Placebo matched to Ivacaftor — Film coated tablet, oral use
  Arms: PC Phase: VX -661 placebo qd + IVA placebo q12h; PC Phase: VX 661 placebo q12h + IVA placebo q12h

SUMMARY:
The objective of this study was to evaluate the safety and efficacy of VX-661in combination with ivacaftor in participants with cystic fibrosis (CF) who are homozygous for F508del cystic fibrosis transmembrane conductance regulator (CFTR) mutation

ELIGIBILITY:
Inclusion Criteria:

* Homozygous for the F508del CFTR mutation
* FEV1 ≥40% and ≤90% of predicted normal for age, sex, and height
* Stable CF disease as judged by the investigator

Exclusion Criteria:

* History of any comorbidity that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant
* Pregnant and nursing females: Females of childbearing potential must have a negative pregnancy test at screening and Day 1 of the PC Phase and Day -7 or Day 1 of the OLE Phase (whichever was applicable)
* Sexually active participants of reproductive potential who are not willing to follow the contraception requirements
* The participant or a close relative of the participant is the investigator or sub investigator, research assistant, pharmacist, study coordinator, or other staff directly involved with the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2016-05-27 (Actual); Study Completion 2016-05-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Birmingham, Alabama
  - Palo Alto, California
  - Stanford, California
  - Altamonte Springs, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Boise, Idaho
  - Chicago, Illinois
  - Boston, Massachusetts
  - New Brunswick, New Jersey
  - New York, New York
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Memphis, Tennessee
  - Houston, Texas
  - Burlington, Vermont
  - Colchester, Vermont
  - Seattle, Washington
  - Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of 2 phases: a randomized, double-blind, placebo-controlled (PC) phase in which participants received either VX-661 in combination with Ivacaftor (IVA), or matched placebo and an open-label extension (OLE) phase in which participants received VX-661 in combination with IVA.
Groups:
- PC Phase: VX-661 50 mg q12h + IVA 150 mg q12h: Participants received VX-661 50 milligram (mg) tablet plus IVA 150 mg tablet every 12 hours (q12h) for 12 weeks.
- PC Phase: VX-661 Placebo q12h + IVA Placebo q12h: Participants received placebo matched to VX-661 tablet plus placebo matched to IVA tablet q12h for 12 weeks.
Period: PC Phase (12 Weeks)
Arm/Group | PC Phase: VX-661 50 mg q12h + IVA 150 mg q12h | PC Phase: VX-661 Placebo q12h + IVA Placebo q12h | PC Phase: VX-661 100 mg qd + IVA 150 mg q12h | PC Phase: VX -661 Placebo qd + IVA Placebo q12h | OLE Phase: VX-661 100 mg qd + IVA 150 mg q12h
Started | 6 | 5 | 15 | 14 | 0
Treated | 6 | 5 | 15 | 13 | 0
Completed | 6 | 5 | 15 | 13 | 0
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — Randomized, but not treated | 0 | 0 | 0 | 1 | 0
Period: OLE Phase (48 Weeks)
Arm/Group | PC Phase: VX-661 50 mg q12h + IVA 150 mg q12h | PC Phase: VX-661 Placebo q12h + IVA Placebo q12h | PC Phase: VX-661 100 mg qd + IVA 150 mg q12h | PC Phase: VX -661 Placebo qd + IVA Placebo q12h | OLE Phase: VX-661 100 mg qd + IVA 150 mg q12h
Started | 0 | 0 | 0 | 0 | 27 (12 participants completed PC phase, but did not enter OLE phase.)
Completed | 0 | 0 | 0 | 0 | 24
Not Completed | 0 | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2
Not completed — Other | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) was defined as all randomized participants who received at least 1 dose of study drug in PC Phase.
Groups:
- PC Phase: VX-661 50 mg q12h + IVA 150 mg q12h: Participants received VX-661 50 mg tablet plus IVA 150 mg tablet q12h for 12 weeks.
- PC Phase: VX-661 100 mg qd + IVA 150 mg q12h: Participants received two VX-661 50 mg tablets qd plus IVA 150 mg tablet q12h for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | PC Phase: VX-661 50 mg q12h + IVA 150 mg q12h | PC Phase: VX-661 Placebo q12h + IVA Placebo q12h | PC Phase: VX-661 100 mg qd + IVA 150 mg q12h | PC Phase: VX -661 Placebo qd + IVA Placebo q12h | Total
Number analyzed (Participants) | 6 | 5 | 15 | 13 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.0 (10.6) | 24.2 (2.2) | 27.3 (5.2) | 30.3 (10.8) | 28.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 7 | 3 | 14
  Male | 4 | 3 | 8 | 10 | 25

OUTCOME MEASURES:

1. Primary Outcome: PC Phase: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: Any untoward medical occurrence in a participant during the study; the event does not necessarily have a causal relationship with the treatment. This includes any newly occurring event or previous condition that has increased in severity or frequency after the informed consent form is signed. AE includes serious as well as Non-serious AEs. SAE (subset of AE): medical event or condition, which falls into any of the following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, Inpatient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event. AEs with start date or increased severity on or after the first dose of study drug through the end of study participation considered treatment-emergent. Baseline was defined as Day 1 of PC Phase.
Time Frame: Baseline (PC Phase) up to 112 days
Population: Safety Set was defined as all participants who received at least 1 dose of study drug in PC Phase.
Measure: Count of Participants; unit: Participants
Arm/Group | PC Phase: VX-661 50 mg q12h + IVA 150 mg q12h | PC Phase: VX-661 Placebo q12h + IVA Placebo q12h | PC Phase: VX-661 100 mg qd + IVA 150 mg q12h | PC Phase: VX -661 Placebo qd + IVA Placebo q12h
Number analyzed (Participants) | 6 | 5 | 15 | 13
Participants
  Participants with AEs | 6 | 5 | 15 | 13
  Participants with SAEs | 1 | 2 | 4 | 5

2. Primary Outcome: OLE Phase: Number of Participants With Treatment-Emergent AEs and SAEs
Description: AE: Any untoward medical occurrence in a participant during the study; the event does not necessarily have a causal relationship with the treatment. This includes any newly occurring event or previous condition that has increased in severity or frequency after the informed consent form is signed. AE includes serious as well as Non-serious AEs. SAE (subset of AE): medical event or condition, which falls into any of the following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, Inpatient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event. AEs with start date or increased severity on or after the first dose of study drug through the end of study participation considered treatment-emergent. Baseline was defined as Day 1 of the OLE Phase.
Time Frame: Baseline (OLE Phase) up to 364 days
Population: Safety Set was defined as all participants who received at least 1 dose of study drug in OLE Phase.
Measure: Count of Participants; unit: Participants
Arm/Group | OLE Phase: VX-661 100 mg qd + IVA 150 mg q12h
Number analyzed (Participants) | 27
Participants
  Participants with AEs | 25
  Participants with SAEs | 6

3. Secondary Outcome: PC Phase: Absolute Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) Through Week 12
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Baseline was defined as Day 1 of PC Phase.
Time Frame: Baseline (PC Phase), Through Week 12
Population: FAS was defined as all randomized participants who received at least 1 dose of study drug in PC Phase.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent predicted of FEV1
Arm/Group | PC Phase: VX-661 50 mg q12h + IVA 150 mg q12h | PC Phase: VX-661 Placebo q12h + IVA Placebo q12h | PC Phase: VX-661 100 mg qd + IVA 150 mg q12h | PC Phase: VX -661 Placebo qd + IVA Placebo q12h
Number analyzed (Participants) | 6 | 5 | 15 | 13
Percent predicted of FEV1 | 0.9 [-3.1 to 5.0] | -0.1 [-4.4 to 4.3] | 3.0 [0.4 to 5.5] | 1.9 [-0.9 to 4.6]

4. Secondary Outcome: OLE Phase: Absolute Change From Baseline in Percent Predicted FEV1 Through Week 40
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Baseline was defined as Day 1 of the OLE Phase.
Time Frame: Baseline (OLE Phase), Through Week 40
Population: Analysis population was defined as all participants who received at least 1 dose of study drug in OLE phase.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent predicted of FEV1
Groups:
- OLE Phase:VX-661 100 mg qd + IVA 150 mg q12h: Participants who completed 12 week PC phase underwent a washout period of at least 4 weeks before entering the OLE phase and received two VX-661 50 mg tablets qd plus IVA 150 mg tablet q12h for 48 weeks in OLE phase.
Arm/Group | OLE Phase:VX-661 100 mg qd + IVA 150 mg q12h
Number analyzed (Participants) | 27
Percent predicted of FEV1 | 2.7 [0.4 to 4.9]

5. Secondary Outcome: PC Phase: Relative Change From Baseline in Percent Predicted FEV1 Through Week 12
Description: as for outcome 3
Time Frame: Baseline (PC Phase), Through Week 12
Population: FAS was defined as all randomized participants who received at least 1 dose of study drug in PC Phase.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Groups:
- PC Phase: VX-661 50 mg + IVA 150 mg: Participants received VX-661 50 mg tablet plus IVA 150 mg tablet q12h for 12 weeks.
Arm/Group | PC Phase: VX-661 50 mg + IVA 150 mg | PC Phase: VX-661 Placebo q12h + IVA Placebo q12h | PC Phase: VX-661 100 mg qd + IVA 150 mg q12h | PC Phase: VX -661 Placebo qd + IVA Placebo q12h
Number analyzed (Participants) | 6 | 5 | 15 | 13
Percent change | 2.6 [-6.0 to 11.1] | 1.0 [-8.2 to 10.3] | 6.0 [0.6 to 11.3] | 4.2 [-1.5 to 10.0]

6. Secondary Outcome: OLE Phase: Relative Change From Baseline in Percent Predicted FEV1 Through Week 40
Description: as for outcome 4
Time Frame: Baseline (OLE Phase), Through Week 40
Population: Analysis population was defined as all participants who received at least 1 dose of study drug in the OLE Phase.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | OLE Phase: VX-661 100 mg qd + IVA 150 mg q12h
Number analyzed (Participants) | 27
Percent change | 6.1 [1.7 to 10.5]

7. Secondary Outcome: PC Phase: Absolute Change From Baseline in Sweat Chloride Through Week 12
Description: Sweat samples were collected using an approved collection device. Baseline was defined as Day 1 of PC Phase.
Time Frame: Baseline (PC Phase), Through Week 12
Population: FAS was defined as all randomized participants who received at least 1 dose of study drug in PC Phase. Here, "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Millimole per liter (mmol/L)
Arm/Group | PC Phase: VX-661 50 mg q12h + IVA 150 mg q12h | PC Phase: VX-661 Placebo q12h + IVA Placebo q12h | PC Phase: VX-661 100 mg qd + IVA 150 mg q12h | PC Phase: VX -661 Placebo qd + IVA Placebo q12h
Number analyzed (Participants) | 5 | 5 | 13 | 13
Millimole per liter (mmol/L) | -10.6 [-16.6 to -4.6] | 2.9 [-3.0 to 8.9] | -4.7 [-8.4 to -0.9] | 0.8 [-3.1 to 4.7]

8. Secondary Outcome: OLE Phase: Absolute Change From Baseline in Sweat Chloride Through Week 40
Description: Sweat samples were collected using an approved collection device. Baseline was defined as Day 1 of the OLE Phase.
Time Frame: Baseline (OLE Phase), Through Week 40
Population: Analysis population was defined as all participants who received at least 1 dose of study drug in the OLE Phase. Here, "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | OLE Phase: VX-661 100 mg qd + IVA 150 mg q12h
Number analyzed (Participants) | 25
mmol/L | -6.6 [-9.7 to -3.5]

9. Secondary Outcome: PC Phase: Absolute Change From Baseline in Body Weight at Week 12
Description: Baseline was defined as Day 1 of PC Phase.
Time Frame: Baseline (PC Phase), Week 12
Population: FAS was defined as all randomized participants who received at least 1 dose of study drug in PC Phase.
Measure: Least Squares Mean (95% Confidence Interval); unit: kilogram (kg)
Arm/Group | PC Phase: VX-661 50 mg q12h + IVA 150 mg q12h | PC Phase: VX-661 Placebo q12h + IVA Placebo q12h | PC Phase: VX-661 100 mg qd + IVA 150 mg q12h | PC Phase: VX -661 Placebo qd + IVA Placebo q12h
Number analyzed (Participants) | 6 | 5 | 15 | 13
kilogram (kg) | 1.0 [-0.4 to 2.3] | 1.6 [0.1 to 3.0] | 0.5 [-0.3 to 1.4] | 0.3 [-0.6 to 1.3]

10. Secondary Outcome: OLE Phase: Absolute Change From Baseline in Body Weight at Week 40
Description: Baseline was defined as Day 1 of the OLE Phase.
Time Frame: Baseline (OLE Phase), Week 40
Population: Analysis population was defined as all participants who received at least 1 dose of study drug in the OLE Phase.
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | OLE Phase: VX-661 100 mg qd + IVA 150 mg q12h
Number analyzed (Participants) | 27
kg | 1.0 [-0.2 to 2.2]

11. Secondary Outcome: PC Phase: Absolute Change From Baseline Body Mass Index (BMI) at Week 12
Description: BMI was calculated using following formula: BMI = Weight in kg/height in square meter (m^2). Baseline was defined as Day 1 of PC Phase.
Time Frame: Baseline (PC Phase), Week 12
Population: FAS was defined as all randomized participants who received at least 1 dose of study drug in PC Phase.
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilogram per square meter (kg/m^2)
Arm/Group | PC Phase: VX-661 50 mg q12h + IVA 150 mg q12h | PC Phase: VX-661 Placebo q12h + IVA Placebo q12h | PC Phase: VX-661 100 mg qd + IVA 150 mg q12h | PC Phase: VX -661 Placebo qd + IVA Placebo q12h
Number analyzed (Participants) | 6 | 5 | 15 | 13
Kilogram per square meter (kg/m^2) | 0.38 [-0.08 to 0.84] | 0.54 [0.03 to 1.04] | 0.18 [-0.11 to 0.47] | 0.11 [-0.21 to 0.42]

12. Secondary Outcome: OLE Phase: Absolute Change From Baseline BMI at Week 40
Description: BMI was calculated using following formula: BMI = Weight in kg/height in m^2. Baseline was defined as Day 1 of the OLE Phase.
Time Frame: Baseline (OLE Phase), Week 40
Population: Analysis population was defined as all participants who received at least 1 dose of study drug in the OLE Phase.
Measure: Least Squares Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | OLE Phase: VX-661 100 mg qd + IVA 150 mg q12h
Number analyzed (Participants) | 27
kg/m^2 | 0.33 [-0.09 to 0.74]

13. Secondary Outcome: PC Phase: Absolute Change From Baseline in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score Through Week 12
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms (for example, coughing, congestion, wheezing), score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life. Baseline was defined as Day 1 of PC Phase.
Time Frame: Baseline (PC Phase), Through Week 12
Population: FAS was defined as all randomized participants who received at least 1 dose of study drug in PC Phase.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PC Phase: VX-661 50 mg q12h + IVA 150 mg q12h | PC Phase: VX-661 Placebo q12h + IVA Placebo q12h | PC Phase: VX-661 100 mg qd + IVA 150 mg q12h | PC Phase: VX -661 Placebo qd + IVA Placebo q12h
Number analyzed (Participants) | 6 | 5 | 15 | 13
units on a scale | 5.6 [-3.9 to 15.1] | -4.6 [-14.9 to 5.7] | 1.0 [-5.1 to 7.0] | 0.4 [-6.2 to 7.1]

14. Secondary Outcome: OLE Phase: Absolute Change From Baseline in CFQ-R Respiratory Domain Score Through Week 40
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms (for example, coughing, congestion, wheezing), score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life. Baseline was defined as Day 1 of the OLE Phase.
Time Frame: Baseline (OLE Phase), Through Week 40
Population: Analysis population was defined as all participants who received at least 1 dose of study drug in the OLE Phase.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | OLE Phase: VX-661 100 mg qd + IVA 150 mg q12h
Number analyzed (Participants) | 27
units on a scale | -0.6 [-5.8 to 4.5]

15. Secondary Outcome: PC Phase: Maximum Plasma Concentration (Cmax) of VX-661 and IVA
Time Frame: Pre-dose, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 85
Population: Analysis population included all participants who received a dose of VX-661 and IVA, whether the participant completed dosing or not and if the dataset(s) supported the noncompartmental analyses.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | PC Phase: VX-661 50 mg q12h + IVA 150 mg q12h | PC Phase: VX-661 100 mg qd + IVA 150 mg q12h
Number analyzed (Participants) | 6 | 15
Nanogram per milliliter (ng/mL)
  VX-661 | 4890 (3150) | 6460 (1240)
  IVA | 1490 (1150) | 1210 (585)

16. Secondary Outcome: PC Phase: Area Under the Concentration Versus Time Curve From Time 0 to 24 Hours (AUC0-24h) of VX-661
Description: Pharmacokinetic (PK) sampling was performed up to 12 hours post-dose on Day 85. For Arm VX-661 50 mg q12h + IVA 150 mg q12h (VX-661 q12h regimen), area under the concentration versus time curve from time 0 to 12 hours (AUC0-12h) was multiplied by 2 to obtain AUC0-24h.
Time Frame: Pre-dose, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 85
Population: Analysis population included all participants who received a dose of VX-661 and IVA, whether the participant completed dosing or not and if the dataset(s) supported the noncompartmental analyses. Here, "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Hour*nanogram per milliliter (hr*ng/mL)
Arm/Group | PC Phase: VX-661 50 mg q12h + IVA 150 mg q12h | PC Phase: VX-661 100 mg qd + IVA 150 mg q12h
Number analyzed (Participants) | 5 | 15
Hour*nanogram per milliliter (hr*ng/mL) | 84900 (55900) | 75500 (20300)

17. Secondary Outcome: PC Phase: Area Under the Concentration Versus Time Curve From Time 0 to 12 Hours (AUC0-12h) of IVA
Time Frame: Pre-dose, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 85
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | PC Phase: VX-661 50 mg q12h + IVA 150 mg q12h | PC Phase: VX-661 100 mg qd + IVA 150 mg q12h
Number analyzed (Participants) | 5 | 15
hr*ng/mL | 14700 (11600) | 10100 (4890)

18. Secondary Outcome: PC Phase: Time to Reach Cmax (Tmax) of VX-661 and IVA
Time Frame: Pre-dose, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 85
Population: as for outcome 15
Measure: Median (Full Range); unit: hour
Arm/Group | PC Phase: VX-661 50 mg q12h + IVA 150 mg q12h | PC Phase: VX-661 100 mg qd + IVA 150 mg q12h
Number analyzed (Participants) | 6 | 15
hour
  VX-661 | 2.48 [1.75 to 4.08] | 3.23 [1.92 to 6.03]
  IVA | 3.59 [1.98 to 6.00] | 4.00 [2.98 to 6.03]

ADVERSE EVENTS:
Time Frame: Baseline (Day 1 of PC Phase) up to 112 days (Placebo control phase); Baseline (Day 1 of OLE Phase) up to 364 days (OLE phase)
Description: Safety Set was defined as all participants who received at least 1 dose of study drug in PC Phase and OLE Phase.
Arm/Group | PC Phase: VX-661 50 mg q12h + IVA 150 mg q12h | PC Phase: VX 661 Placebo q12h + IVA Placebo q12h | PC Phase: VX-661 100 mg qd + IVA 150 mg q12h | PC Phase: VX -661 Placebo qd + IVA Placebo q12h | OLE Phase: VX-661 100 mg qd + IVA 150 mg q12h
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 0/15 | 0/13 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/6 | 2/5 | 4/15 | 5/13 | 6/27
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5 | 15/15 | 13/13 | 25/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PC Phase: VX-661 50 mg q12h + IVA 150 mg q12h (N=6) | PC Phase: VX 661 Placebo q12h + IVA Placebo q12h (N=5) | PC Phase: VX-661 100 mg qd + IVA 150 mg q12h (N=15) | PC Phase: VX -661 Placebo qd + IVA Placebo q12h (N=13) | OLE Phase: VX-661 100 mg qd + IVA 150 mg q12h (N=27)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 2 | 4 | 4 | 5
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Cystic fibrosis related diabetes (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PC Phase: VX-661 50 mg q12h + IVA 150 mg q12h (N=6) | PC Phase: VX 661 Placebo q12h + IVA Placebo q12h (N=5) | PC Phase: VX-661 100 mg qd + IVA 150 mg q12h (N=15) | PC Phase: VX -661 Placebo qd + IVA Placebo q12h (N=13) | OLE Phase: VX-661 100 mg qd + IVA 150 mg q12h (N=27)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 4 | 5 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 1 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 3 | 3
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 3 | 2
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 2 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 3
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary function test decreased (Investigations) | 1 | 1 | 2 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 2 | 1 | 3
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 2
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 1 | 0
Heart rate increased (Investigations) | 0 | 1 | 1 | 0 | 0
Blood bilirubin unconjugated increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 1 | 0 | 0
Breath sounds abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Urine output decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Forced expiratory volume decreased (Investigations) | 0 | 1 | 0 | 2 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 0 | 2 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0
Vitamin A decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Vitamin K decreased (Investigations) | 0 | 0 | 0 | 1 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 1 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 | 3 | 5 | 4 | 13
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 2
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 3 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2
Headache (Nervous system disorders) | 1 | 0 | 2 | 1 | 4
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Hyposmia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 1 | 0 | 2
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0
Vaccination site discomfort (General disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Vitamin E deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.